CLINICAL TRIAL: NCT00917228
Title: A Wireless Lingual Feedback Device to Reduce Overpressures in Seated Posture: A Feasibility Study
Acronym: prevesc0001
Status: Completed | Type: Observational
Sponsor: TIMC-IMAG (Other)
Collaborators: Olivier Chenu (Unknown); Nicolas Vuillerme (Unknown); Jacques Demongeot (Unknown); Yohan Payan (Unknown)
Other Study IDs: prevesc0001
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Postural Behaviour; Overpressures Reductions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Feedback: Subjects of this group are equipped with the biofeedback system
  Interventions: Device: recordings with device equipped
- Control: Subjects of this group are not equipped with the biofeedback system
  Interventions: Device: Control

INTERVENTIONS:
Device: recordings with device equipped
  Groups: Feedback
Device: Control — Recording without device equipped
  Groups: Control

SUMMARY:
This study evaluates the feasibility of a biofeedback system aimed at reducing overpressures during seated posture. The system consists of (1) a pressure sensors map, (2) a laptop that couples sensors with actuators, (3) a Tongue Display Unit (TDU) consisting of a wireless circuit embedded in a dental retainer with a matrix of electrodes. The principle of this biofeedback system consists in (1) detecting overpressures in people who are seated over long periods of time, (2) estimating a postural change that could reduce these overpressures and (3) communicating this change through directional information transmitted by the TDU.

It is hypothesized that overpressures are diminished after biofeedback.

ELIGIBILITY:
Inclusion Criteria:

* young healthy subjects

Exclusion Criteria:

* motor or sensory disabilities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy subjects
Sampling Method: Non-Probability Sample

PRIMARY OUTCOMES:
Ability to reach a target posture | 10 seconds
Decrease of the overpressures at the seat/body interface | 10 seconds
Decrease of overpressures bigger for higher pressures | 10 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Timc-Imag, La Tronche, France